CLINICAL TRIAL: NCT04209803
Title: Efficacy and Tolerability of N-Acetyl- Cysteine for Treatment of The Early-onset Androgenetic Alopecia in Men
Brief Title: N-Acetyl-Cysteine for Treatment of AGA in Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Aboshabana Hussein Mohamed, Teaching Assistant of Dermatology and Venereology Department Kafrelsheikh University, Kafrelsheikh University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: N-Acetyl- Cysteine for AGA
Record Dates: First submitted 2019-12-12; First posted 2019-12-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Minoxidil group (Active Comparator): The first group will receive Minoxidil 5% topically twice daily for 4 months.
  Interventions: Drug: Minoxidil 5% topically and oral NAC 600 mg
- NAC group (Active Comparator): The second group will receive NAC orally 600 mg 3 times a day for 4 months.
  Interventions: Drug: Minoxidil 5% topically and oral NAC 600 mg
- Minoxidil + NAC group (Active Comparator): The third group will receive combined treatment of Minoxidil 5% twice daily and oral NAC 600 mg 3 times a day for 4 months.
  Interventions: Drug: Minoxidil 5% topically and oral NAC 600 mg
- Control group (No Intervention): The fourth group will be the patients who are refusing the treatment and will be followed-up over 4 months.

INTERVENTIONS:
Drug: Minoxidil 5% topically and oral NAC 600 mg — Topical 5% Minoxidil and N-Acetyl-Cysteine 600 mg orally
  Other Names: Hair Back scalp lotion 5% and Acetylcistein 600 mg sachet
  Arms: Minoxidil + NAC group; Minoxidil group; NAC group

SUMMARY:
To study the effectiveness and safety of the reactive oxygen species scavenger N-acetyl-cysteine (NAC) as a single therapy and in combination with the topically applied minoxidil for the treatment of the early-onset androgenetic alopecia in men.

DETAILED DESCRIPTION:
Androgenetic alopecia (AGA) is a non-scarring disease with a progressive thinning of the scalp hair that follows a characteristic pattern. AGA, the most common form of hair loss in men, involves the progressive loss of visible pigmented terminal hair on the scalp in response to circulating androgens. AGA is an autosomal disorder that begins in puberty in genetically predisposed individuals. Thinning usually begins between the age of 12 and 40 years in both sexes, and at least 50% of the men by the age of 50 and 50% of women by 60 years are more affected. The pathogenesis of androgenetic alopecia involves both genetic and hormonal factors. The hair follicles are genetically targeted for androgen stimulation leading to follicular miniaturization and replacement of large pigmented hairs (terminal hairs) with shorter, thinner depigmented hairs (vellus hairs) in affected areas. Environmental factors, the nutritional influences, metabolic syndrome, smoking, and UV radiation, also play a role in the pathogenesis of AGA. Recent histological studies illustrated perifollicular inflammation in the upper third of the hair follicles, suggesting that inflammation plays a pathogenic role in AGA, although clinically, AGA is considered a non-inflammatory disease. Oxidative stress and inflammation are closely linked in biological systems. The enhanced hair loss in androgenetic alopecia was linked to several factors that increase cellular oxidative stress, including metabolic syndrome, alcohol consumption, smoking, and UV radiation. AGA patients were found to suffer from oxidative stress as evidenced by the decreased total antioxidant activity as well as increased malondialdehyde levels. Erdogan et al.investigated the oxidative stress in early-onset androgenetic alopecia and found that the total oxidant levels and oxidative stress index are higher in younger patients with early-onset AGA. Molecular studies of the paracrine mediators around the dermal papilla cells have shed light on the role played by ROS in bald scalp. Prostaglandin D2 (PGD2) was found to be elevated in the bald scalp of AGA patients and negatively affected the growth of human hair. PGD2 was found to enhance the capacity of human keratinocytes to convert the weak androgen, androstenedione, to testosterone through the involvement of the ROS cellular signaling axis. The ROS scavenger, N-acetyl-cysteine, blocked the enhanced testosterone production by PGD2. Transforming growth factor-beta (TGF-β) is another key promotor of hair follicle apoptosis. TGF-β was found to be androgen-inducible via the induction of ROS and its induction was significantly suppressed by the ROS-scavenger, N-acetyl cysteine in the hair follicle dermal papilla cells. Treatment of cases of androgenetic alopecia comprises a therapeutic challenge. AGA is neither life-threatening nor does it lead to pain; however, it leads to a significant emotional burden and is considered as a therapeutically frustrating disorder to the patients. The therapeutic approach to the patient with androgenetic alopecia should be global: combined treatments may obtain improvements in hair density, reduction of miniaturization and hair loss. Minoxidil 2% or 5% solution is the most frequently used drug for topical application. In men with AGA, 5% topical minoxidil was clearly superior to 2% topical minoxidil in increasing hair regrowth.

Men who used 5% topical minoxidil also had an earlier response to treatment than those who used 2% topical minoxidil. Psychosocial perceptions of hair loss in men with AGA were also improved. Finasteride, a selective inhibitor of 5α- reductase of type II reduces the conversion of testosterone into DHT, was approved by FDA in 1997 in a dosage of 1 mg/day as a systemic therapy in adult men with mild to moderate AGA. N-acetylcysteine (NAC) has been widely used as an antioxidant in vivo and in vitro. N-Acetylcysteine may act as a precursor of glutathione facilitating its biosynthesis. Glutathione will then serve as a protective agent and detoxify reactive species both enzymatically and non-enzymatically. It is possible that N-acetylcysteine could scavenge the active oxygen species directly by non-enzymatic reduction. By replenishing glutathione, NAC can prevent paracetamol toxicity. NAC is traditionally used as a hepatoprotective agent for the treatment of paracetamol toxicity. Its mucolytic and anti-inflammatory actions allow its successful use in chronic bronchopulmonary disease. Dermatologically, NAC in a dose ranging from 1200 mg/day up to 2400 mg/day constitutes an effective treatment of trichotillomania owing to its glutamate modulating action via the reduction of oxidative stress and normalization of glutaminergic transmission. It is generally well tolerated with a high safety profile, mild gastrointestinal symptoms like vomiting and diarrhea are the most common side effects. Given that oxidative stress emerges as a new component in the multifactorial milieu of the aetiopathogenesis of AGA; the proved high oxidative stress index in patients with early-onset androgenetic alopecia; the established in vitro efficacy of ROSscavenger, N-acetyl cysteine, in blocking ROS and subsequently the inhibitory paracrine mediators (PGD2 & TGF-β) of the hair follicle dermal papilla in the bald scalp; together with the high safety profile and tolerability of NAC, the investigators thought to investigate the efficacy and tolerability of NAC as a single therapy and in combination with minoxidil for treatment of the early-onset androgenetic alopecia in men.

ELIGIBILITY:
Inclusion Criteria:

* Male patients between 18-30 years old affected by mild to moderate AGA up to grade IV on the Norwood-Hamilton scale.

Exclusion Criteria:

* Patients with contraindication to intake of NAC like patients on nitrates.
* Patients with AGA who were on systemic treatment (Finasteride, Dutasteride) in the previous 12 months.
* Patients with AGA who received topical treatment for AGA in the last 6 months.
* Patients with AGA taking any antioxidants, food and vitamin supplements within the last 3 months.
* Patients with pathological systemic diseases or environmental factors which provide a high oxidative stress state including heavy smoking, alcohol consumption, diagnosis of metabolic syndrome, and prolonged exposure to ultraviolet.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Assessment by digital images for effectiveness | 4 months
  A photographic review of the scalp for each patient. Photos were standardized as to subject, area, distance, illumination, angle of exposure and background so that there were no major differences between any of the series of photographs. Photographs were taken using Nikon D3300 AF-P 18-55 VR 24.2 Megapixels® digital camera, based on the grading suggested by Olsen et al.,(2002) graded the photographs on a 7-point scale from dense, moderate, minimal growth, no change, minimal, moderate or dense loss. This was shown at baseline and 16 weeks of the trial.
Trichoscopic assessment for effectiveness | 4 months
  Images were taken from fixed points in the scalp using the Dermlite П PRO HR® dermoscopy for each patient when they first presented and every month for four months. Digital images of the dermoscopic features were taken by digital camera Nikon D3300 AF-P 18-55 VR 24.2 Megapixels®. The reference points are set to the top of the vertex and a landmark for each frontal region was the intersecting point between lines passing through the ipsilateral tragus and lateral point of eyebrows. Each point was analyzed before and after follow up period by single-blinded expert in trichoscopy looking for the following parameters; total hair count, terminal hair count, vellus hair count, triple or more follicular unit, double follicular unit, single follicular unit, number of perifollicular halo (peripilar sign), thick terminal hair and thin terminal (intermediate) hair. Parameters recorded numerically then statistically analyzed for comparison between different groups of trial.
Patient satisfaction towards treatment outcome. | 4 months
  Patient satisfaction scaled from 0 if unsatisfied, 1 is mild satisfied and 2 if satisfied and compliance with treatment was documented through a patient-filled questionnaire.
Side effects towards treatment used in trial. | 4 months
  Side effects of the drugs (irritation, dandruff, and hypertrichosis for minoxidil plus nausea for NAC) were documented and statistically analyzed for comparison between groups of trial.

CONTACTS AND LOCATIONS:
Overall Officials: Mahira H El Sayed, Professor, Study Chair — Ain Shams University- Faculty of Medicine
Locations (1):
- dermatology clinics in Ain Shams University Hospital and Kafr El Sheik University Hospital., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaya Erdogan H, Bulur I, Kocaturk E, Yildiz B, Saracoglu ZN, Alatas O. The role of oxidative stress in early-onset androgenetic alopecia. J Cosmet Dermatol. 2017 Dec;16(4):527-530. doi: 10.1111/jocd.12300. Epub 2016 Dec 16. PMID 27987270
- [Background] Mantel A, McDonald JT, Goldsborough K, Harvey VM, Chan J. Prostaglandin D2 Uses Components of ROS Signaling to Enhance Testosterone Production in Keratinocytes. J Investig Dermatol Symp Proc. 2017 Oct;18(2):S81-S84. doi: 10.1016/j.jisp.2017.01.003. PMID 28941500
- [Background] Barroso LAL, Sternberg F, Souza MNIFE, Nunes GJB. Trichotillomania: a good response to treatment with N-acetylcysteine. An Bras Dermatol. 2017 Jul-Aug;92(4):537-539. doi: 10.1590/abd1806-4841.20175435. PMID 28954106